CLINICAL TRIAL: NCT05761236
Title: The Effect of Pilates-Based Exercises Practised by Hybrid Telerehabilitation on Respiratory Functions, Respiratory Muscle Strength and Functional Capacity
Brief Title: Pilates-Based Exercises Practised by Hybrid Telerehabilitation in Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ayşe Sena Manzak, Research Asssistant, Bezmialem Vakif University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BVUaysesena02
Record Dates: First submitted 2023-02-02; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Pilates; Telerehabilitation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Active Comparator): In the first 2 weeks, sessions were held with all patients once a week. In these two sessions, the basic information of scoliosis were explained to both groups. Postural corrections were explained to the patients, including the basic elements of clinical pilates.It was stated that they should breathe towards the concave side of the major curve (weak breathing zone) during exercises and postural corrections.In the Pilates-based exercise program, sessions are planned as 10 minutes of warm-up, 10 minutes of cool-down and 40 minutes of scoliosis-specific pilates-based exercises for approximately 1 hour. Total number of exercises is 12 for one session. After a 2-week joint training week, the training group switched to hybrid type telerehabilitation and continued their exercise sessions with a physiotherapist 3 days a week via synchronous video conferences (Zoom Application) and by themselves at home on the rest of the week.
  Interventions: Other: Exercise
- Control group (Active Comparator): In the first 2 weeks, sessions were held with all patients once a week. In these two sessions, the basic information of scoliosis were explained to both groups. Postural corrections were explained to the patients, including the basic elements of clinical pilates. It was stated that they should breathe towards the concave side of the major curve (weak breathing zone) during exercises and postural corrections.In the Pilates-based exercise program, sessions are planned as 10 minutes of warm-up, 10 minutes of cool-down and 40 minutes of scoliosis-specific pilates-based exercises for approximately 1 hour. Total number of exercises is 12 for one session.The patients in the control group continued the exercise program every day of the week for 12 weeks. Exercise lists were sent to the patients in the form of electronic booklets via an electronic communication application every week, and their continuity with the exercise program was checked with the diaries they were asked to fill in.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Sessions are consisted of scoliosis-specific pilates-based exercises.The exercises were kept constant in total content, but the bilateral or unilateral application directions, the number of repetitions for the right and left sides, and the extremities used were modified for each patient according to the localization of the major curve and the type of the curve. The taught postural corrections were requested to be maintained during all exercises. Exercises for flexibility were performed asymmetrically or symmetrically according to the chosen exercise, extremities were chosen according to the curve type, with 5 repetitions and 30 seconds for each repetition. Exercises aimed at strengthening were performed for a total of 12 repetitions, during a 5-second contraction, by arranging the number of repetitions for the right and left in line with the target muscles, again considering the curve type, and the patients were asked to rest between the exercises.

SUMMARY:
The aim of this study was to see the effect of pilates-based exercise training applied with hybrid telerehabilitation method on Cobb angle, trunk rotation angle (ATR), respiratory functions, respiratory muscle strength and functional capacity in children with AIS between the ages of 10-18 and home-based pilates exercise. compare its effectiveness with respect to its training. Investigators of this study think that synchronous telerehabilitation sessions added to home-based pilates exercise training in children with AIS with moderate and moderate-to-severe curves can have positive effects on the evaluation parameters examined, and the results of this study can guide the relevant physiotherapists and health professionals by adding a new perspective to the literature.

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) is defined as a deformity characterized by abnormal spinal curve formation and rotation of the vertebrae in the coronal plane in a healthy individual aged 10 years and older, without any known cause.This study aimed to investigate the effect of pilates-based exercise training applied with hybrid telerehabilitation method on Cobb angle, respiratory function, respiratory muscle strength and functional capacity in patients with AIS, including postural corrections and breathing pattern determined by curve type-localization. Within the scope of the study, 32 patients diagnosed with AIS, aged 10-18 years, were randomized and divided into education and control groups. Cobb angle measurement, trunk rotation angle measurement, respiratory function test, respiratory muscle strength, functional capacity were evaluated in all patients. Training and control groups participated in supervised sessions once a week during the first 2 weeks of exercise training processes. During these sessions, the patients were informed about the basics of pilates, the postural corrections determined according to the curve type and localization, and the respiratory principles. For the next 10 weeks, the training group took synchronous online sessions with a physiotherapist 3 days a week, and the exercises were continued at home for 4 days. The control group, on the other hand, continued the same exercises 7 days a week, home-based for 10 weeks. At the end of 12 weeks, all assessments were repeated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIS between the ages of 10-18
* Cobb angle is between 25-50 degrees
* Desktop-laptop computers, smart phones, electronic tablets, etc., which will provide internet connection and video-conferencing facilities in the homes of the patients
* The child is not included in another treatment program that will affect the progression of scoliosis

Exclusion Criteria:

* Surgical operation in the last 3 months
* The child has a neurological, orthopedic or systemic disease that will prevent him from exercising
* Having communicative, cognitive and behavioral disorders that may cause problems in understanding commands and questions during assessment and exercises
* Exercising regularly at least 3 days a week

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Cobb angle | 12 weeks
  When measuring the Cobb angle, the tangent lines on the radiological film are drawn from the superior end plate of the superior vertebra participating in the curvature and the inferior endplate of the lowest vertebra participating in the curvature. The angle formed at the intersection of these two lines is the Cobb angle. The evaluation was performed by the same physician before and after the treatment.
Pulmonary function | 12 weeks
  Spirometry device was used in the evaluation of lung functions and measurements were carried out in accordance with ATS/ERS criteria. Before the test, the weight, height, age and gender values of the patients were recorded on the spirometer device. All of the measurements were made in the sitting position with the feet in full contact with the ground. A nose clip was used. At the beginning of the test, inspiration and expiration were requested at the tidal volume limits. Afterwards, rapid expiration was requested following the deepest possible inspiration. Care was taken to maintain the expiration time for 6 seconds without interruption. It was recorded by choosing the best of three tests that were 95% consistent with each other. Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), Tiffeneau ratio (FEV1/FVC) and peak expiratory volume (PEF) values were measured and both measured values and percentages of expected values were recorded.
Respiratory muscle strength | 12 weeks
  Respiratory muscle strength was measured in accordance with ATS/ERS criteria using an electronic and portable intraoral pressure measuring device.All of the measurements were made in the sitting position with the feet in full contact with the ground. Nasal breathing was blocked with a nose clip. In order to measure the maximum inspiratory pressure (MIP), maximum expiratory maneuver was performed before the patient took the mouthpiece of the device into his mouth, and then maximal inspiration (Müller maneuver) was performed at maximum speed for 1-3 seconds. For maximum expiratory pressure measurement, the maximum inspiratory maneuver was performed before the mouthpiece of the device was taken into the mouth, and then maximal expiration (Valsalva maneuver) was performed at maximum speed for 1-3 seconds. 3 measurements were repeated for each evaluation and the highest value was recorded in "cmH2O".
Functional capacity | 12 weeks
  ISWT is a test consisting of 12 levels and each level lasts 1 minute.In ISWT the walking area was arranged to be 10 meters for each shuttle. By observing the signals heard between the two cones; patients walked very slowly at first, then at an increasing speed with 3 beeps at the end of each minute. The test was terminated in cases where the test could not be continued or if a signal was received when 0.5 m or more from the cones twice consecutively. In ESWT test, peak oxygen consumption was calculated and the value corresponding to 85% of the peak VO2 was placed on the graph and the velocity was found. After the first 2-minute warm-up period of the test, the patients were asked to walk with the determined speed. In cases where the test could not be continued, the test was terminated if the signal was received 0.5 m or more from the cones twice consecutively, and if the maximum test time of 20 minutes was reached. Walking time was recorded in seconds.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bezmialem Vakıf University, Istanbul, Eyüp
  - Bezmialem Vakıf University, Istanbul

REFERENCES:
- [Derived] Manzak Dursun AS, Ozyilmaz S, Ucgun H, Elmadag NM. The effect of Pilates-based exercise applied with hybrid telerehabilitation method in children with adolescent idiopathic scoliosis: A randomized clinical trial. Eur J Pediatr. 2024 Feb;183(2):759-767. doi: 10.1007/s00431-023-05340-2. Epub 2023 Nov 23. PMID 37993666